CLINICAL TRIAL: NCT00993655
Title: A Phase II Study of Intraperitoneal (IP) Plus Intravenous (IV) Chemotherapy Versus IV Carboplatin Plus Paclitaxel in Patients With Epithelial Ovarian Cancer Optimally Debulked at Surgery Following Neoadjuvant Intravenous Chemotherapy
Brief Title: Intraperitoneal vs Intravenous Chemotherapy Following Neoadjuvant Chemotherapy in Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Grupo Español de Investigación en Cáncer de Ovario (Other); Cancer Research UK (Other); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OV21; CAN-NCIC-OV21 (Registry Identifier: PDQ (NCI US Physician Data Query)); UCL08/0379 (Other: NCI); GEICO-0902 (Other: GEICO); SWOG OV.21 (Other: South West Oncology Group); CDR0000655241 (Other: PDQ)
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2020-03

CONDITIONS: Fallopian Tube Cancer; Metastatic Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: peritoneal cavity cancer; fallopian tube cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; malignant pleural effusion; ovarian clear cell cystadenocarcinoma; ovarian clear cell tumor with proliferating activity
MeSH Terms: conditions — Fallopian Tube Neoplasms; Neoplasm Metastasis; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Pleural Effusion, Malignant | interventions — Carboplatin; Cisplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- IV carboplatin + IV paclitaxel (Active Comparator): ARM 1: Paclitaxel 135 mg/m2 intravenous day 1 plus Carboplatin AUC 5 if measured GFR or AUC6 if estimated GFR intravenous day 1; Paclitaxel 60 mg/m2 intravenous day 8. Cycles given Q 21 days x 3 cycles
  Interventions: Drug: carboplatin; Drug: paclitaxel
- IP cisplatin + IV/IP paclitaxel (Active Comparator): ARM 2: Paclitaxel 135 mg/m2 intravenous day 1 plus Cisplatin 75 mg/m2 intraperitoneal day 1; Paclitaxel 60 mg/m2 intraperitoneal day 8. Cycles given Q 21 days x 3 cycles (Phase II cisplatin arm closed to accrual on 2014-FEB-03)
  Interventions: Drug: cisplatin; Drug: paclitaxel
- IP carboplatin + IV/IP paclitaxel (Active Comparator): ARM 3: Paclitaxel 135 mg/m2 intravenous day 1 plus Carboplatin AUC 5 if measured GFR or AUC6 if estimated GFR intraperitoneal day 1; Paclitaxel 60 mg/m2 intraperitoneal day 8. Cycles given Q 21 days x 3 cycles
  Interventions: Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: carboplatin — Carboplatin AUC 5 if measured GFR or AUC6 if calculated GFR intravenous or intraperitoneal.
  Arms: IP carboplatin + IV/IP paclitaxel; IV carboplatin + IV paclitaxel
Drug: cisplatin — Cisplatin 75 mg/m2 intraperitoneal day 1
  Arms: IP cisplatin + IV/IP paclitaxel
Drug: paclitaxel — Paclitaxel 135 mg/m2 intravenous day 1 plus Paclitaxel 60 mg/m2 intraperitoneal or intravenously day 8. Cycles given Q 21 days x 3 cycles

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, carboplatin, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) and giving them in different ways may kill more tumor cells. It is not yet known which combination chemotherapy regimen is more effective in treating patients with ovarian epithelial cancer, primary peritoneal cancer, and fallopian tube cancer.

PURPOSE: This randomized phase II trial is comparing the side effects of three combination chemotherapy regimens and to see how well they work in treating patients with stage IIB, stage IIC, stage III, or stage IV ovarian epithelial cancer, primary peritoneal cancer, or fallopian tube cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the efficacy of the selected IP chemotherapy regimen (Arm 3: IV paclitaxel and IP carboplatin plus day 8 IP paclitaxel) versus IV carboplatin plus paclitaxel (Arm 1) in patients with epithelial ovarian cancer optimally debulked at surgery following neoadjuvant intravenous chemotherapy. Nine month progressive rate post randomization is the primary endpoint for assessment of efficacy.

Secondary

* To compare IP plus IV chemotherapy versus IV carboplatin plus paclitaxel with respect to progression free survival and overall survival.

OUTLINE: This is a multicenter study. Patients are stratified according to cooperative group, residual disease (observable [e.g., macroscopic] disease that is evident at end of delayed primary debulking surgery vs no evidence of observable disease at end of delayed primary debulking surgery), reason for delayed primary debulking surgery at initial diagnosis (nonresectable disease vs other reasons), and timing of intraperitoneal catheter insertion (intra-operative catheter insertion vs post-operative insertion).

* Phase II: Patients are randomized to 1 of 3 treatment groups.

  * ARM 1: Paclitaxel 135 mg/m2 intravenous day 1 plus Carboplatin AUC 5 if measured GFR or AUC6 if estimated GFR intravenous day 1; Paclitaxel 60 mg/m2 intravenous day 8. Cycles given Q 21 days x 3 cycles
  * ARM 2: Paclitaxel 135 mg/m2 intravenous day 1 plus Cisplatin 75 mg/m2 intraperitoneal day 1; Paclitaxel 60 mg/m2 intraperitoneal day 8. Cycles given Q 21 days x 3 cycles (Phase II cisplatin arm closed to accrual on 2014-Feb-03)
  * ARM 3: Paclitaxel 135 mg/m2 intravenous day 1 plus Carboplatin AUC 5 if measured GFR or AUC6 if estimated GFR intraperitoneal day 1; Paclitaxel 60 mg/m2 intraperitoneal day 8. Cycles given Q 21 days x 3 cycles.

Patients also receive carboplatin IP on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity.

* Expanded Phase II: Patients are randomized to 1 of 2 treatment groups.

  * Arm I: Patients receive paclitaxel and carboplatin as in phase II, arm I.
  * Arm III: Patients receive paclitaxel and cisplatin as in phase II, arm II or paclitaxel and carboplatin as in phase II, arm III.

Patients complete quality of life questionnaires EORTC QLQ-C30, ovarian cancer module (EORTC QLQ-OV28), and FACT/GOG-Ntx at baseline, on day 1 of courses 2 and 3, at 3, 6 and 12 months after completion of study treatment, and then annually until disease progression, death, or initiation of second-line therapy.

After completion of study treatment, patients are followed at 6 weeks, every 3 months for 2 years, every 6 months for 2 years, and then annually until progression, death, or initiation of second-line therapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, primary serous type peritoneal, or fallopian tube carcinoma

  * Patients with ovarian cancer of the clear cell histology are eligible. Histologic confirmation is preferably by biopsy or limited excision prior to neo-adjuvant treatment. If the diagnosis prior to neo-adjuvant chemotherapy is based on cytology, histologic confirmation is required prior to randomization. Histologic confirmation can be obtained at the time of debulking surgery by intra-operative frozen section, thus permitting intra-operative randomization, or by final pathologic review of the resected specimen if randomization is to be performed following debulking surgery.
  * Initial FIGO stage IIB-III disease

    * Stage IV disease allowed provided the only criterion for stage IV disease is the presence of a pleural effusion confirmed to be associated with positive cytology for ovarian cancer
* Completed ≥ 3 but no more than 4 courses of platinum-based neoadjuvant chemotherapy prior to the first debulking surgery
* Meets the following criteria for surgical treatment prior to randomization:

  * Initial Diagnosis: No debulking surgery was attempted or completed.
  * The patient's first cytoreductive (debulking) surgery must be after neoadjuvant chemotherapy (Delayed Primary Debulking). The delayed primary debulking surgery must be completed no more than 4 weeks after commencing administering of the last cycle of neoadjuvant chemotherapy and must be completed no more than 6 weeks prior to randomization.
  * Surgery will include total abdominal hysterectomy, bilateral salpingo-oophorectomy, omentectomy and any additional procedures required to achieve maximal cytoreduction with residual disease of 1 cm or less as assessed by the surgeon at the end of surgery.

    * Delayed primary debulking surgery must be completed no more than 4 weeks after the last course of neoadjuvant chemotherapy and must be completed no more than 6 weeks prior to randomization
  * Surgery will include total abdominal hysterectomy, bilateral salpingo-oophorectomy, omentectomy, and any additional procedures required to achieve maximal cytoreduction with residual disease of ≤ 1 cm as assessed by the surgeon at the end of surgery
* No borderline ovarian tumors (i.e., tumors of low malignant potential) alone
* No mucinous tumor

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Granulocyte count ≥ 1.5 x 10^9/L
* Platelet count ≥ 100 x 10^9/L
* Serum creatinine ≤ upper limit of normal (ULN) OR > ULN to ≤ 1.25 ULN provided measured creatinine clearance is > 60 mL/min
* Serum bilirubin normal
* AST/ALT ≤ 2.5 times ULN
* Fertile patients must use effective contraception
* Able (i.e., sufficiently fluent) and willing to complete the quality of life questionnaires
* Accessible for treatment and follow-up
* No history of other malignancy, except adequately treated nonmelanoma skin cancer, curatively treated carcinoma in situ of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years
* No uncontrolled atrial or ventricular arrhythmias including second or third degree heart block unless managed with implanted pacemaker

  * Patients with a history of first degree heart block are eligible
* No documented myocardial infarction within the past 6 months preceding randomization (pretreatment ECG evidence only of infarct will not exclude patients)
* No diagnosis of bowel obstruction
* No serious illness or medical condition which would not permit the patient to be managed according to protocol including, but not limited to, any of the following:

  * Prior allergic reactions to drugs containing cremophor or to compounds chemically related to cisplatin, paclitaxel, or carboplatin
  * Symptomatic congestive heart failure within the past 6 months or other conditions which would lead to a contraindication of a high-volume saline diuresis
  * History of significant neurologic or psychiatric disorder which would impair the ability to obtain consent
  * Active uncontrolled infection
  * Persistent peripheral neuropathy or hearing loss ≥ grade 2 resulting from prior therapy
  * Extensive intraperitoneal adhesion intra- or post-operatively which would impede intraperitoneal treatment delivery

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior therapy for ovarian cancer, except for neoadjuvant platinum-based chemotherapy and surgery
* No concurrent intraperitoneal adhesion barriers
* No other concurrent anticancer treatment, including cytotoxic agents, biological response modifiers, immunotherapy, anticancer hormone therapy, or investigational drug therapy
* No other concurrent experimental drugs or anticancer therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2010-03-03 (Actual); Primary Completion 2016-03-10 (Actual); Study Completion 2016-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen J. Mackay, MD, Study Chair — Princess Margaret Hospital, Canada; Diane M. Provencher, MD, FRCS, FACOG, Study Chair — Hopital Notre-Dame du CHUM
Locations (50):
- United States (6):
  - Mercy-Springfield, Springfield, Missouri
  - CoxHealth, Springfield, Missouri
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Univ of Utah (Huntsman Cancer Institute), Salt Lake City, Utah
  - Northwest CCOP - Multicare Health System, Tacoma, Washington
- Canada (19):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Regional Health Authority B, Zone 2, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
- Spain (10):
  - Instituto Catalan de Oncologia - L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Fundacion Alcorcon, Alcorcón, Madrid
  - Hospital Vall d'Hebron, Barcelona
  - Corporacio Sanitaria Clinic, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Gregorio Maranon, Madrid
  - Centro Oncologico MD Anderson - Madrid, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Fundacion Instituto Valenciano de Oncologia, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (15):
  - The Clatterbridge Center for Oncology - Liverpool, Metropolitan Borough of Wirral, Bebington
  - Mount Vernon Hospital - Middlesex, Middlesex, Northwood
  - St. George's Hospital - London, London, Tooting
  - Wexham Park Hospital, Slough, Wexham
  - The Christie Hospital - Manchester, Manchester, Withington
  - The Western General Hospital - Edinburgh, Edinburgh
  - St. James University Hospital - Leeds, Leeds
  - Liverpool Women's Hospital - Liverpool, Liverpool
  - St. Bartholomew's Hospital - London, London
  - The Royal Marsden Hospital - London, London
  - The Hammersmith Hospital - London, London
  - University College London Hospital - London, London
  - St Marys Hospital - Manchester, Manchester
  - The Churchill Hospital - Oxford, Oxford
  - The Derriford Hospital - Plymouth, Plymouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Provencher DM, Gallagher CJ, Parulekar WR, Ledermann JA, Armstrong DK, Brundage M, Gourley C, Romero I, Gonzalez-Martin A, Feeney M, Bessette P, Hall M, Weberpals JI, Hall G, Lau SK, Gauthier P, Fung-Kee-Fung M, Eisenhauer EA, Winch C, Tu D, MacKay HJ. OV21/PETROC: a randomized Gynecologic Cancer Intergroup phase II study of intraperitoneal versus intravenous chemotherapy following neoadjuvant chemotherapy and optimal debulking surgery in epithelial ovarian cancer. Ann Oncol. 2018 Feb 1;29(2):431-438. doi: 10.1093/annonc/mdx754. PMID 29186319

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: ARM 1: Paclitaxel 135 mg/m2 intravenous day 1 plus Carboplatin AUC 5 if measured GFR or AUC6 if estimated GFR intravenous day 1; Paclitaxel 60 mg/m2 intravenous day 8. Cycles given Q 21 days x 3 cycles
  carboplatin: Carboplatin AUC 5 if measured GFR or AUC6 if calculated GFR intravenous or intraperitoneal.
  paclitaxel: Paclitaxel 135 mg/m2 intravenous day 1 plus Paclitaxel 60 mg/m2 intraperitoneal or intravenously day 8. Cycles given Q 21 days x 3 cycles
- Arm 2: ARM 2: Paclitaxel 135 mg/m2 intravenous day 1 plus Cisplatin 75 mg/m2 intraperitoneal day 1; Paclitaxel 60 mg/m2 intraperitoneal day 8. Cycles given Q 21 days x 3 cycles (Phase II cisplatin arm closed to accrual on 2014-FEB-03)
  cisplatin: Cisplatin 75 mg/m2 intraperitoneal day 1
  paclitaxel: Paclitaxel 135 mg/m2 intravenous day 1 plus Paclitaxel 60 mg/m2 intraperitoneal or intravenously day 8. Cycles given Q 21 days x 3 cycles
  quality-of-life assessment: day 1 cycle 2, day 1 cycle 3 and at 3, 6, 12 mo then annually until disease progression, death or initiation of second-line therapy
- Arm 3: ARM 3: Paclitaxel 135 mg/m2 intravenous day 1 plus Carboplatin AUC 5 if measured GFR or AUC6 if estimated GFR intraperitoneal day 1; Paclitaxel 60 mg/m2 intraperitoneal day 8. Cycles given Q 21 days x 3 cycles
  paclitaxel: Paclitaxel 135 mg/m2 intravenous day 1 plus Paclitaxel 60 mg/m2 intraperitoneal or intravenously day 8. Cycles given Q 21 days x 3 cycles
  quality-of-life assessment: day 1 cycle 2, day 1 cycle 3 and at 3, 6, 12 mo then annually until disease progression, death or initiation of second-line therapy
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3
Started | 101 | 72 | 102
Completed | 101 | 72 | 102
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Total
Number analyzed (Participants) | 101 | 72 | 102 | 275
Age, Continuous [Median (Full Range); unit: years] | 62 [33 to 83] | 61 [29 to 78] | 62 [40 to 82] | 62 [29 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 72 | 102 | 275
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 5 | 1 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 1 | 3
  Black or African American | 1 | 1 | 1 | 3
  White | 92 | 67 | 95 | 254
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 65 | 42 | 66 | 173
  United States | 3 | 4 | 3 | 10
  United Kingdom | 27 | 20 | 27 | 74
  Spain | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: 9-month Progression Rate Post-randomization
Description: It is defined as proportion of patients who had progressed at or before 9 months after randomization, i.e., the time from the randomization to the date when the first observation of disease progression (earliest of the date when the first CA 125 meets progression definition and the date of first objective relapse or progression, defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions, recorded) has been documented or when death due to any cause has been observed was less than or equal to 9 months.
Time Frame: 9 months
Population: All randomized patients
Measure: Number; unit: Porportion of participants
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 101 | 72 | 102
Porportion of participants | 0.386 | 0.347 | 0.245
Statistical Analysis 1: Comparison: Arm 1 vs Arm 3; Assume that the 9-month PD rate in IV arm (Arm 1) will be 40% (based on experience with data from NCIC CTG OV.16 and that of NCRI UK). The target sample size of 200 will enable the detection of a 19% difference between Arms 1 and 3 in 9 month progression disease rate post randomization with 80% power at two-sided 0.05 level; Test type: Superiority; p = 0.065, Cochran-Mantel-Haenszel; adjusting for stratification factors at randomization

2. Secondary Outcome: Progression Free Survival
Description: Time from the day of randomization until the time when first observation of disease progression (earliest of the dates of first CA125 which meets progression definition and first objective relapse or progression defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions, has been documented or when death due to any cause has been observed.
Time Frame: During the study with median follow-up of 33 months
Population: All patients randomized to the study
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IV Carboplatin + IV Paclitaxel | IP Cisplatin + IV/IP Paclitaxel | IP Carboplatin + IV/IP Paclitaxel
Number analyzed (Participants) | 101 | 72 | 102
months | 11.3 [8.8 to 14.7] | 12.7 [9.7 to 18.0] | 12.5 [10.8 to 15.0]
Statistical Analysis 1: Comparison: IV Carboplatin + IV Paclitaxel vs IP Carboplatin + IV/IP Paclitaxel; Test type: Superiority; p = 0.27, Log Rank; Adjusting for stratification factors at randomization; Hazard Ratio (HR) = 1.22, 95% CI 2-sided [0.85 to 1.75]

3. Secondary Outcome: Overall Survival
Description: Time from the day of randomization to death from any cause.
Time Frame: During the study with median follow-up of 33 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IV Carboplatin + IV Paclitaxel | IP Cisplatin + IV/IP Paclitaxel | IP Carboplatin + IV/IP Paclitaxel
Number analyzed (Participants) | 101 | 72 | 102
months | 38.1 [32.9 to 47.7] | 40.6 [38.7 to 68.1] | 59.3 [34.2 to 68.3]
Statistical Analysis 1: Comparison: IV Carboplatin + IV Paclitaxel vs IP Carboplatin + IV/IP Paclitaxel; Test type: Superiority; p = 0.40, Log Rank; Adjusting for stratification factors at randomization; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [0.74 to 2.13]

ADVERSE EVENTS:
Time Frame: During the time when patients were treated by protocol therapy, up to 9 months
Arm/Group | Arm 1 | Arm 2 | Arm 3
All-Cause Mortality (participants affected / at risk) | 34/95 | 24/67 | 26/92
Serious Adverse Events (participants affected / at risk) | 7/95 | 8/67 | 6/92
Other Adverse Events (participants affected / at risk) | 94/95 | 64/67 | 92/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=95) | Arm 2 (N=67) | Arm 3 (N=92)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Infusion site extravasation (General disorders) | 0 | 2 | 0
Abdominal infection (Infections and infestations) | 0 | 1 | 0
Pelvic infection (Infections and infestations) | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Infusion related reaction (General disorders) | 0 | 0 | 1
Intraoperative gastrointestinal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=95) | Arm 2 (N=67) | Arm 3 (N=92)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 1 | 1
Palpitations (Cardiac disorders) | 6 | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 7 | 3 | 4
Tinnitus (Ear and labyrinth disorders) | 5 | 11 | 8
Blurred vision (Eye disorders) | 5 | 3 | 5
Abdominal pain (Gastrointestinal disorders) | 45 | 43 | 56
Bloating (Gastrointestinal disorders) | 8 | 15 | 17
Constipation (Gastrointestinal disorders) | 51 | 41 | 54
Diarrhea (Gastrointestinal disorders) | 28 | 19 | 27
Dyspepsia (Gastrointestinal disorders) | 10 | 13 | 6
Gastroesophageal reflux disease (Gastrointestinal disorders) | 12 | 4 | 6
Mucositis oral (Gastrointestinal disorders) | 19 | 5 | 14
Nausea (Gastrointestinal disorders) | 46 | 38 | 51
Vomiting (Gastrointestinal disorders) | 20 | 12 | 20
ther gastrointestinal disorders (Gastrointestinal disorders) | 5 | 4 | 4
Edema limbs (General disorders) | 7 | 7 | 8
Fatigue (General disorders) | 77 | 51 | 72
Pain (General disorders) | 18 | 11 | 11
Anorexia (Metabolism and nutrition disorders) | 22 | 18 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 10 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 10 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 19 | 13 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 | 5 | 11
Dizziness (Nervous system disorders) | 6 | 8 | 10
Dysgeusia (Nervous system disorders) | 14 | 4 | 11
Headache (Nervous system disorders) | 12 | 7 | 10
Paresthesia (Nervous system disorders) | 12 | 7 | 15
Peripheral sensory neuropathy (Nervous system disorders) | 52 | 31 | 43
Anxiety (Psychiatric disorders) | 17 | 11 | 15
Depression (Psychiatric disorders) | 6 | 4 | 4
Insomnia (Psychiatric disorders) | 30 | 20 | 31
Urinary incontinence (Renal and urinary disorders) | 6 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 6 | 8 | 5
Vaginal discharge (Reproductive system and breast disorders) | 6 | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 22 | 8 | 22
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 5
Alopecia (Respiratory, thoracic and mediastinal disorders) | 52 | 35 | 58
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 2 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 6 | 2 | 2
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 8 | 2 | 9
Flushing (Vascular disorders) | 2 | 7 | 6
Hot flashes/ flushes (Vascular disorders) | 17 | 10 | 11
Hypertension (Vascular disorders) | 9 | 5 | 6
Abdominal distension (Gastrointestinal disorders) | 2 | 10 | 6
Flatulence (Gastrointestinal disorders) | 3 | 4 | 5
Infusion site extravasation (General disorders) | 2 | 5 | 2
Other general disorders, administration site conditions (General disorders) | 4 | 6 | 6
Dehydration (Metabolism and nutrition disorders) | 2 | 4 | 0
Urinary frequency (Renal and urinary disorders) | 2 | 5 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 4 | 7
Other surgical and medical procedures (Surgical and medical procedures) | 0 | 5 | 4
Urinary tract infection (Renal and urinary disorders) | 0 | 0 | 5
Other nervous system disorders (Nervous system disorders) | 2 | 0 | 5
Thromboembolic event (Vascular disorders) | 4 | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No